CLINICAL TRIAL: NCT04166591
Title: Learning New Words From Overhearing in Children With ASD
Brief Title: Study 1 Replication and Extension of Prior Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Emerson College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 280521
Record Dates: First submitted 2019-10-31; First posted 2019-11-18 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Addressed (Experimental): Children participate in an interaction with an experimenter who uses the word to be learned.
  Interventions: Behavioral: Addressed Speech
- Overheard (Experimental): Children observe while an experimenter uses the word to be learned in an interaction with another experimenter.
  Interventions: Behavioral: Overheard Speech

INTERVENTIONS:
Behavioral: Overheard Speech — New words are introduced with the child as an observer rather directly taught.
  Arms: Overheard
Behavioral: Addressed Speech — New words are introduced directly to the child by an experimenter.
  Arms: Addressed

SUMMARY:
The goal of this research is to explore abilities to learn word meanings from overheard conversations in children with ASD (and, as a control, typically developing children).

Specific Aim 1 (Experiment 1): Subaim 1a: Identify child characteristics associated with learning from overhearing. In a prior study, the investigators found that 13 children with ASD were able to learn the meanings of novel words that they heard used in a conversation involving two adults. In the current study, the investigators aim to study a larger sample to identify what child characteristics are associated with good learning in an overhearing situation as compared to a situation in which the child is directly taught the new word. Subaim 1b: Assess retention and generalization of words learned from overhearing. The investigators will re-test children on their knowledge of the word meanings after a 10-minute delay to see if they both retain the word meanings and can generalize the new words to new situations.

ELIGIBILITY:
Inclusion Criteria:

* children with or without a diagnosis of ASD between 18 to 71 months of age

Exclusion Criteria:

* native language is not English
* born premature (< 36 weeks)
* has uncorrected hearing or vision impairments
* has developmental disorders or medical conditions other than ASD that affect language or cognition (excepting psychiatric conditions often comorbid with ASD such as ADHD)
* has a history of photosensitive epileptic seizures

Ages: 18 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 342 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Emerson College, Boston, Massachusetts
  - New York University, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ASD - Addressed First, Then Overheard: Children with ASD are exposed to new words.
  Addressed Speech: New words are introduced directly to the child by an experimenter.
  Overheard Speech: New words are introduced while children observe.
- ASD - Overheard First, Then Addressed: Children with ASD are exposed to new words.
  Overheard Speech: New words are introduced while children observe.
  Addressed Speech: New words are introduced directly to the child by an experimenter.
- TD - Addressed First, Then Overheard: Children with TD are exposed to new words.
  Addressed Speech: New words are introduced directly to the child by an experimenter.
  Overheard Speech: New words are introduced while children observe.
- TD - Overheard First, Then Addressed: Children with TD are exposed to new words.
  Overheard Speech: New words are introduced while children observe.
  Addressed Speech: New words are introduced directly to the child by an experimenter.
Period: First Behavioral Task (3 Minutes)
Arm/Group | ASD - Addressed First, Then Overheard | ASD - Overheard First, Then Addressed | TD - Addressed First, Then Overheard | TD - Overheard First, Then Addressed
Started | 87 | 89 | 85 | 81
Completed | 78 | 78 | 83 | 79
Not Completed | 9 | 11 | 2 | 2
Not completed — Withdrawal by Subject | 9 | 11 | 2 | 2
Period: Second Behavioral Task (3 Minutes)
Arm/Group | ASD - Addressed First, Then Overheard | ASD - Overheard First, Then Addressed | TD - Addressed First, Then Overheard | TD - Overheard First, Then Addressed
Started | 87 | 89 | 85 | 81
Completed | 78 | 78 | 83 | 79
Not Completed | 9 | 11 | 2 | 2
Not completed — Withdrawal by Subject | 9 | 11 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASD - Addressed First, Then Overheard | ASD - Overheard First, Then Addressed | TD - Addressed First, Then Overheard | TD - Overheard First, Then Addressed | Total
Number analyzed (Participants) | 87 | 89 | 85 | 81 | 342
Age, Continuous [Mean (Standard Deviation); unit: months] | 51.8 (10.6) | 52.1 (10.2) | 41.5 (14.2) | 31.0 (8.2) | 41.7 (14.3)
Sex/Gender, Customized [Number; unit: participants]
  Number of Enrolled Males | 66 | 66 | 47 | 56 | 235
  Number of Enrolled Females | 21 | 22 | 38 | 25 | 106
  Number Prefer not to Answer | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian / Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 4 | 5 | 4 | 3 | 16
  Black | 10 | 5 | 6 | 4 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  White | 42 | 57 | 52 | 56 | 207
  More than one | 16 | 5 | 17 | 14 | 52
  Unknown | 8 | 14 | 2 | 2 | 26
  Hispanic/Latine | 7 | 3 | 2 | 2 | 14
Region of Enrollment [Number; unit: participants]
  United States | 87 | 89 | 85 | 81 | 342

OUTCOME MEASURES:

1. Primary Outcome: Number of Children Who Select the Target Object as Measured by Gaze Preference.
Description: Children are prompted to identify the object that is associated with the target word.
Time Frame: immediately after viewing 3-minute interaction
Population: Order of conditions, which was counterbalanced in the experimental design, is collapsed for the purposes of analysis. Not all enrolled participants were analyzed because of exclusions due to, e.g., experimenter error or children paying insufficient attention.
Measure: Count of Participants; unit: Participants
Groups:
- ASD - Addressed: Children with ASD are exposed to new words.
  Addressed Speech: New words are introduced directly to the child by an experimenter.
- ASD - Overheard: Children with ASD are exposed to new words.
  Overheard Speech: New words are introduced while children observe.
- TD - Addressed: Children with TD are exposed to new words.
  Addressed Speech: New words are introduced directly to the child by an experimenter.
- TD - Overheard: Children with TD are exposed to new words.
  Overheard Speech: New words are introduced while children observe.
Arm/Group | ASD - Addressed | ASD - Overheard | TD - Addressed | TD - Overheard
Number analyzed (Participants) | 80 | 82 | 106 | 104
Participants | 47 | 44 | 71 | 56
Statistical Analysis 1: Comparison: ASD - Addressed; Test type: Other — The primary statistical analysis involves asking whether children look at the target significantly more than chance levels. Binomial tests are used to see if the number of children who do so is significantly greater than would be expected by chance; p < 0.01, binomial test
Statistical Analysis 2: Comparison: ASD - Overheard; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.01, Binomial test
Statistical Analysis 3: Comparison: TD - Addressed; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.01, Binomial test
Statistical Analysis 4: Comparison: TD - Overheard; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.01, Binomial test

2. Primary Outcome: Number of Children Who Select the Target Object as Measured by Gaze Preference.
Description: Children are prompted to identify the object that is associated with the target word.
Time Frame: 5 minutes after viewing interaction
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- ASD - Addressed; TD - Addressed: Children participate in an interaction with an experimenter who uses the word to be learned.
  Addressed Speech: New words are introduced directly to the child by an experimenter.
- ASD - Overheard; TD - Overheard: Children observe while an experimenter uses the word to be learned in an interaction with another experimenter.
  Overheard Speech: New words are introduced with the child as an observer rather directly taught.
Arm/Group | ASD - Addressed | ASD - Overheard | TD - Addressed | TD - Overheard
Number analyzed (Participants) | 73 | 77 | 98 | 92
Participants | 44 | 31 | 54 | 58
Statistical Analysis 1: Comparison: ASD - Addressed; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.01, Binomial test
Statistical Analysis 2: Comparison: ASD - Overheard; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.12, Binomial test
Statistical Analysis 3: Comparison: TD - Addressed; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.01, Binomial test
Statistical Analysis 4: Comparison: TD - Overheard; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.01, Binomial test

ADVERSE EVENTS:
Time Frame: the duration of study participation (approximately 10 minutes)
Description: Our experimental paradigm involves presenting children with videos of everyday child-friendly actions during a 10-minute interaction. There is no risk of Serious Adverse Events or All-Cause Mortality during the session.
Arm/Group | ASD - Addressed | ASD - Overheard | TD - Addressed | TD - Overheard
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/176 | 0/166 | 0/166
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/176 | 0/166 | 0/166
Other Adverse Events (participants affected / at risk) | 0/176 | 0/176 | 0/166 | 0/166

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT04166591/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT04166591/ICF_000.pdf